CLINICAL TRIAL: NCT00395083
Title: CSP #560 - Bronchitis and Emphysema Advice and Training to Reduce Hospitalization (BREATH)
Brief Title: Bronchitis and Emphysema Advice and Training to Reduce Hospitalization
Acronym: BREATH
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The DMC detected an imbalance in safety outcomes between the two groups.
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 560
Record Dates: First submitted 2006-11-01; First posted 2006-11-02 (Estimated); Results first posted 2014-08-21 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: COPD; Emphysema
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (No Intervention): Patients allocated to the control arm will receive standardized care that incorporates guide-line based recommendations including influenza vaccination, a short-acting bronchodilator, and either a long-acting bronchodilator or inhaled corticosteroid inhaler.
- Group 2 (Experimental): The comprehensive group will receive an initial, intense education program with development of an action plan, and regular telephone contacts by a case manager in addition to standardized COPD care.
  Interventions: Behavioral: COPD Self-management Education

INTERVENTIONS:
Behavioral: COPD Self-management Education — The comprehensive self-management intervention incorporates self-management education, development of an action plan, and case management. The intervention is designed using the social cognitive theory with the Precede-Proceed Model which has guided other successful patient education programs.
  Arms: Group 2

SUMMARY:
EXECUTIVE SUMMARY:

Purpose: To evaluate the efficacy and cost-effectiveness of a novel intervention incorporating self-management education, an action plan, and case-management to decrease the risk of hospitalizations due to chronic obstructive pulmonary disease (COPD) among veterans with severe COPD.

Hypotheses:

Primary Hypothesis:

Veterans with COPD who receive a self-management program incorporating education sessions, development of an action plan, and case-management will have a decreased risk of COPD hospitalization compared to standardized COPD care.

Primary Objective:

In an intent-to-treat analysis, determine the efficacy of a comprehensive self-management program for reducing the risk of COPD hospitalization in veterans with severe COPD in comparison to patients receiving standardized COPD care.

Secondary Hypotheses:

Compared with standardized COPD care, veterans with COPD who receive a comprehensive self-management intervention will have: A) decreased health-related costs resulting from decreased hospitalizations and outpatient utilization, B) decreased hospitalization rates and average length of stay due to both COPD and all-cause admissions, and C) improvement in a set of outcomes including mortality, health-related quality of life, medication adherence, patient satisfaction, disease knowledge, skill acquisition and self-efficacy.

Secondary Objectives:

To evaluate the healthcare costs, hospitalization days, mortality, adherence, and health outcomes of a comprehensive self-management program compared to standardized COPD care among patients with severe COPD measured by:

A)Healthcare-related costs B)Health services use due to COPD and to all causes C)Clinical outcome measures

1. Mortality
2. Health-related quality of life measured by generic and COPD-specific measures
3. Patient satisfaction
4. Medication adherence
5. Disease knowledge, skill acquisition and self-efficacy

In the proposed study, 960 veterans with severe COPD hospitalized in the previous year will be randomly assigned to either a comprehensive case management program or standardized COPD care. The comprehensive group will receive an initial, intense education program with development of an action plan, and regular telephone contacts by a case manager in addition to standardized COPD care. Patients allocated to the control arm will receive standardized care that incorporates guideline-based recommendations including influenza vaccination, a short-acting bronchodilator, and either a long-acting bronchodilator or inhaled corticosteroid inhaler.

The study will be conducted in 2 phases, a 12-month feasibility study conducted at 6 VA sites followed by the full study in which an additional 8 sites will enroll patients over the next 24 months. As a result, 180 patients will be initially enrolled in the feasibility study over the first year and the remaining 780 patients will be enrolled in the second and third years of the study when the full study is implemented. Subjects will be followed until the completion of the study, for at least one, and up to four years. The primary outcome is time to first COPD hospitalization.

DETAILED DESCRIPTION:
EXECUTIVE SUMMARY:

Purpose: To evaluate the efficacy and cost-effectiveness of a novel intervention incorporating self-management education, an action plan, and case-management to decrease the risk of hospitalizations due to chronic obstructive pulmonary disease (COPD) among veterans with severe COPD.

Hypotheses:

Primary Hypothesis:

Veterans with COPD who receive a self-management program incorporating education sessions, development of an action plan, and case-management will have a decreased risk of COPD hospitalization compared to standardized COPD care.

Primary Objective:

In an intent-to-treat analysis, determine the efficacy of a comprehensive self-management program for reducing the risk of COPD hospitalization in veterans with severe COPD in comparison to patients receiving standardized COPD care.

Secondary Hypotheses:

Compared with standardized COPD care, veterans with COPD who receive a comprehensive self-management intervention will have: A) decreased health-related costs resulting from decreased hospitalizations and outpatient utilization, B) decreased hospitalization rates and average length of stay due to both COPD and all-cause admissions, and C) improvement in a set of outcomes including mortality, health-related quality of life, medication adherence, patient satisfaction, disease knowledge, skill acquisition and self-efficacy.

Secondary Objectives:

To evaluate the healthcare costs, hospitalization days, mortality, adherence, and health outcomes of a comprehensive self-management program compared to standardized COPD care among patients with severe COPD measured by:

A)Healthcare-related costs B)Health services use due to COPD and to all causes C)Clinical outcome measures

1. Mortality
2. Health-related quality of life measured by generic and COPD-specific measures
3. Patient satisfaction
4. Medication adherence
5. Disease knowledge, skill acquisition and self-efficacy

In the proposed study, 960 veterans with severe COPD hospitalized in the previous year will be randomly assigned to either a comprehensive case management program or standardized COPD care. The comprehensive group will receive an initial, intense education program with development of an action plan, and regular telephone contacts by a case manager in addition to standardized COPD care. Patients allocated to the control arm will receive standardized care that incorporates guideline-based recommendations including influenza vaccination, a short-acting bronchodilator, and either a long-acting bronchodilator or inhaled corticosteroid inhaler.

The study will be conducted in 2 phases, a 12-month feasibility study conducted at 6 VA sites followed by the full study in which an additional 8 sites will enroll patients over the next 24 months. As a result, 180 patients will be initially enrolled in the feasibility study over the first year and the remaining 780 patients will be enrolled in the second and third years of the study when the full study is implemented. Subjects will be followed until the completion of the study, for at least one, and up to four years. The primary outcome is time to first COPD hospitalization.

Exacerbations among patients with COPD result in costly emergency room visits and hospitalizations. The overall direct and indirect medical costs of COPD for the United States in 2000 were estimated to be in excess of $30 billion. In the VA health care system, there were 16,073 discharges for COPD in fiscal year 2003 at an average cost of $9,400 (2005 dollars). Disease management programs for COPD may improve patient self-care, improving symptoms and resulting in decreased exacerbations. However, implementing the types of published programs that use self-management education and case-management require additional resources for the VA. The COPD disease management program described in this proposal was developed by extensive modification of existing programs using the strongest theory-based and evidence-based elements, and takes advantage of existing VA systems. By targeting patients at high risk for exacerbations, this study focuses on the population in which the needs and potential impact are the greatest.

The intervention is designed to enable patients with COPD to manage their disease more effectively, by monitoring their symptoms and initiating appropriate action when their symptoms worsen. The elements of the program are developed using self-efficacy theory, a recognized and powerful predictor of health-related behavior change. The goal of the intervention is an informed and activated patient working with an informed, skilled case manager to improve self-management of COPD and ultimately clinical outcomes. Case-management programs are used to improve outcomes and to reduce health care utilization among patients with other chronic diseases such as diabetes, congestive heart failure and asthma, suggesting that this approach may be successful in COPD.

A study conducted in Canada by Dr. Bourbeau, a co-investigator for this proposal, suggests that an intensive home-based self-management education program and case-management reduce the risk of COPD hospitalizations by 35% over 1-year, and reduced average hospital days by 42%. Cost-savings resulting from decreased hospitalizations offset the cost of the intervention, and the intervention was potentially cost-saving. Relying on home visits, the intervention is not practical or affordable in the VA, and therefore this study evaluates whether a novel case-management intervention for COPD developed specifically for the VA will reduce hospitalizations without increasing overall health-care costs.

Because the majority of health care costs for patients with COPD are due to hospitalizations for exacerbations, COPD admissions are the primary outcome and the principal self-management goal. Assessing the cost-effectiveness of this intervention is a critical component of the proposed study, and will provide data for evidence-based decisions by VA physicians and managers regarding the management of COPD.

ELIGIBILITY:
Inclusion Criteria:

Population to be studied

The study population consists of VA patients with COPD who receive some of their medical care at Veterans Affairs medical centers and were hospitalized for COPD in the last 12 months. To ensure that patients enrolled in the study receive regular care at the participating VA, we will include only patients enrolled in either the primary care or pulmonary clinic at the VA medical center and were seen at least once in the last year. This criterion should not significantly decrease the number of eligible patients because 90% of patients admitted for COPD in the VA had at least 1 outpatient visit to the VA primary care clinic in the year prior to their hospitalization based on data from the VA OPC in FY03.

Inclusion Criteria:

1. Diagnosis of COPD confirmed by all of the following:

   1. FEV1/FVC < 0.70
   2. FEV1 < 80%
   3. Age > 40 years
   4. A current or past history of cigarette smoking (> 10 pack-years)
2. COPD hospitalization in the previous year
3. Receives care at participating VA medical center

   1. Enrolled in either primary care or pulmonary clinic at the VA
   2. Seen at least once in the past year in either primary care or pulmonary clinic
4. No COPD exacerbations in last 4 weeks
5. English-speaking
6. Access to telephone

Exclusion Criteria:

1. Primary clinical diagnosis of asthma
2. Medical conditions affecting the ability to participate in the study such as:

   1. Comorbid illness likely to limit life expectancy < 1 year
   2. Decompensated heart failure
   3. Dementia
   4. Uncontrolled psychiatric illness
3. Participation in another clinical intervention trial in the previous 30 days

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 426 (Actual)
Dates: Start 2006-07; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent S. Fan, MD MPH, Study Chair — VA Puget Sound Health Care System
Locations (22):
- United States (22):
  - Carl T. Hayden VA Medical Center, Phoenix, Arizona
  - Southern Arizona VA Health Care System, Tucson, Tucson, Arizona
  - VA Medical Center, Loma Linda, Loma Linda, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - VA Medical Center, Bay Pines, Bay Pines, Florida
  - North Florida/South Georgia Veterans Health System, Gainesville, Florida
  - Atlanta VA Medical and Rehab Center, Decatur, Decatur, Georgia
  - Richard Roudebush VA Medical Center, Indianapolis, Indianapolis, Indiana
  - Robert J. Dole VAMC & ROC, Wichita, Wichita, Kansas
  - VA Medical Center, Lexington, Lexington, Kentucky
  - VA Medical Center, Kansas City MO, Kansas City, Missouri
  - New Mexico VA Health Care System, Albuquerque, Albuquerque, New Mexico
  - VA Western New York Healthcare System at Buffalo, Buffalo, New York
  - New York Harbor HCS, New York, New York
  - VA Medical Center, Cincinnati, Cincinnati, Ohio
  - VA Medical Center, Oklahoma City, Oklahoma City, Oklahoma
  - VA Medical Center, Providence, Providence, Rhode Island
  - VA North Texas Health Care System, Dallas, Dallas, Texas
  - Michael E. DeBakey VA Medical Center (152), Houston, Texas
  - VA South Texas Health Care System, San Antonio, San Antonio, Texas
  - Hunter Holmes McGuire VA Medical Center, Richmond, Virginia
  - VA Puget Sound Health Care System, Seattle, Washington

REFERENCES:
- [Result] Fan VS, Gaziano JM, Lew R, Bourbeau J, Adams SG, Leatherman S, Thwin SS, Huang GD, Robbins R, Sriram PS, Sharafkhaneh A, Mador MJ, Sarosi G, Panos RJ, Rastogi P, Wagner TH, Mazzuca SA, Shannon C, Colling C, Liang MH, Stoller JK, Fiore L, Niewoehner DE. A comprehensive care management program to prevent chronic obstructive pulmonary disease hospitalizations: a randomized, controlled trial. Ann Intern Med. 2012 May 15;156(10):673-83. doi: 10.7326/0003-4819-156-10-201205150-00003. PMID 22586006

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The pilot study began in July 2006, and trial recruitment began in January 2007 with 6 sites, later expanding to 20. Recruitment ended early in March 2009 due to DMC recommendations.
Groups:
- Usual Care: Patients allocated to the control arm will receive standardized care that incorporates guide-line based recommendations including influenza vaccination, a short-acting bronchodilator, and either a long-acting bronchodilator or inhaled corticosteroid inhaler.
- Comprehensive Care Management Program: The comprehensive group will receive an initial, intense education program with development of an action plan, and regular telephone contacts by a case manager in addition to standardized COPD care.
  COPD Self-management Education: The comprehensive self-management intervention incorporates self-management education, development of an action plan, and case management. The intervention is designed using the social cognitive theory with the Precede-Proceed Model which has guided other successful patient education programs.
Period: Overall Study
Arm/Group | Usual Care | Comprehensive Care Management Program
Started | 217 | 209
Completed | 207 | 201
Not Completed | 10 | 8
Not completed — Withdrawal by Subject | 6 | 5
Not completed — Developed another disease | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Comprehensive Care Management Program | Total
Number analyzed (Participants) | 217 | 209 | 426
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (8.2) | 66.2 (8.4) | 66.0 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 209 | 204 | 413
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 3 | 8
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 20 | 24 | 44
  White | 191 | 181 | 372
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 2 | 10
  Not Hispanic or Latino | 209 | 207 | 416
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Hospitalization-free Survival - Time to Event
Time Frame: From randomization until date of first hospitalization for COPD, assessed up to 26 months
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Usual Care | Comprehensive Care Management Program
Number analyzed (Participants) | 217 | 209
years | 0.45 [0.36 to 0.53] | 0.46 [0.39 to 0.54]
Statistical Analysis 1: Comparison: Usual Care vs Comprehensive Care Management Program; Test type: Superiority or Other; p = 0.62, Log Rank; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.70 to 1.80]

2. Primary Outcome: Hazard Ratio for First COPD Hospitalization
Time Frame: 26 months
Measure: Number; unit: participants
Arm/Group | Usual Care | Comprehensive Care Management Program
Number analyzed (Participants) | 217 | 209
participants
  Subjects with COPD Hospitalization | 34 | 36
  Subjects without COPD Hospitalization | 183 | 173
Statistical Analysis 1: Comparison: Usual Care vs Comprehensive Care Management Program; Test type: Superiority or Other; p = 0.62, Regression, Cox; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.70 to 1.80]

3. Secondary Outcome: Hazard Ratio for All-Cause Mortality
Time Frame: 26 months
Measure: Number; unit: participants
Arm/Group | Usual Care | Comprehensive Care Management Program
Number analyzed (Participants) | 217 | 209
participants
  All-Cause Death | 10 | 28
  Alive | 207 | 181
Statistical Analysis 1: Comparison: Usual Care vs Comprehensive Care Management Program; Test type: Superiority or Other; p = 0.003, Regression, Cox; Hazard Ratio (HR) = 3.00, 95% CI 2-sided [1.46 to 6.17]

4. Secondary Outcome: Time to All-Cause Death
Time Frame: From randomization until death, assessed up to 26 months
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Usual Care | Comprehensive Care Management Program
Number analyzed (Participants) | 217 | 209
years | 0.51 [0.43 to 0.79] | 0.49 [0.40 to 0.61]
Statistical Analysis 1: Comparison: Usual Care vs Comprehensive Care Management Program; Test type: Superiority or Other; p = 0.002, Log Rank; Hazard Ratio (HR) = 3.00, 95% CI 2-sided [1.46 to 6.17]

ADVERSE EVENTS:
Description: Non-serious adverse events were not collected for this study.
Arm/Group | Usual Care | Comprehensive Care Management Program
Serious Adverse Events (participants affected / at risk) | 98/217 | 91/209
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=217) | Comprehensive Care Management Program (N=209)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Angina pectoris (Cardiac disorders) | 2 (2) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 2 (5)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 8 (12)
Myocardial infarction (Cardiac disorders) | 4 (4) | 3 (3)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 3 (4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal infarction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Volvulus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Adverse drug reaction (General disorders) | 2 (2) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 7 (7) | 4 (4)
Death (General disorders) | 3 (3) | 6 (6)
Fatigue (General disorders) | 1 (1) | 0 (0)
Hernia (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2) | 2 (3)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 2 (2)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Infective exacerbation of chronic obstructive (Infections and infestations) | 1 (1) | 0 (0)
Lung infection pseudomonal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 17 (19) | 17 (21)
Prostate infection (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection staphylococal (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 3 (4)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Biopsy lung (Investigations) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1)
Tuberculin test positive (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Aggression (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Drug abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0)
Bladder mass (Renal and urinary disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 2 (2) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 53 (84) | 42 (65)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 4 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Physical assault (Social circumstances) | 0 (0) | 1 (2)
Angioplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Bladder operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Carotid endarterectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Colectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Hospitalisation (Surgical and medical procedures) | 1 (1) | 0 (0)
Implantable defibrillator insertion (Surgical and medical procedures) | 1 (1) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Palliative care (Surgical and medical procedures) | 0 (0) | 1 (1)
Preoperative care (Surgical and medical procedures) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 0 (0) | 3 (3)
Aortic aneurysm rupture (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 1 (2) | 0 (0)
Subclavian artery stenosis (Vascular disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
Hepatitis alcoholic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Alocholism (Psychiatric disorders) | 1 (2) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes